CLINICAL TRIAL: NCT00921583
Title: Long-term Examination of Titanium Dental Implants With a TPS Surface: A Prospective 20-year Case Series Study
Status: Completed | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Chappuis Vivianne, Dep. of Oral Surgery and Stomatology, University of Bern
Other Study IDs: KEK 078/09
Record Dates: First submitted 2009-05-28; First posted 2009-06-16 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Dental Implants; Periimplantitis
Keywords: survival rate; success rate
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Examination of dental implants 20 years in function
  Interventions: Device: Long-term examination

INTERVENTIONS:
Device: Long-term examination — Follow-up dental implants 20 year in function

SUMMARY:
Since 1986, newly developed titanium implants with a TPS surface have been utilized for the treatment of partially edentulous patients with implant supported fixed dental prostheses (FTP). In the beginning, these implant types have been sold by Straumann under the brand name "Bonefit implants", later "ITI Dental Implant System" From the beginning, the first 75 patients have been documented in a prospective case series study, and clinical and radiographic results have been reported at 1-year, 3-years, 5-years and 8-years.

The aim of the present study is to examine the long-term outcomes of this original group of patients with at 20 years of clinical function, and to assess the frequency of biological and technical complications during this follow-up period.

DETAILED DESCRIPTION:
Background:

The rehabilitation with implant-supported restorations has been a successful treatment modality in fully and partially edentulous patients since the early 1980s . Today, partially edentulous individuals have become the main group of patients being considered for implant therapy, and several reports have been published showing favorable long-term outcomes with different dental implant systems. In systematic reviews analyzing the long-term performance of osseointegrated implants, clinical studies with 5-year observation periods are frequently included. However, studies with a 10-year observation period are sparse. Only three clinical studies with an observation period of 20-years in edentulous or partially edentulous patients have been found.

Objective:

The objective is to evaluate dental implants after 20 years of function.

Methods:

Partially edentulous patients provided with implants between 1986 and 1989 at the Department of Oral Surgery and Stomatology at the University of Bern recruited for a clinical and radiographic evaluation 20 years after implant installation. A total of 75 patients with 102 implants will be recalled for a clinical and radiographic examination. All implants installed were hollow screw and hollow cylinder implants (Straumann, Waldenburg, Switzerland) with a rough TPS surface. They were placed according to the manufacturer's guidelines. The superstructures consistent in single crowns or fixed partial dentures, which were incorporated 4-6 months postsurgically. All patients will be evaluated using information from patient's charts and from the 20-year examination. Apical radiographs will be taken from the implant and the adjacent tooth. The marginal bone level around the adjacent tooth will also be calculated using the implant shoulder a reference point.

ELIGIBILITY:
Inclusion Criteria:

* Original group of patient

Exclusion Criteria:

* Other patient than from original group

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Partially edentulous patients provided with implants between 1986 and 1989 at the Department of Oral Surgery and Stomatology at the University of Bern recruited for a clinical and radiographic evaluation 20 years after implant installation. A total of 75 patients with 102 implants will be recalled for a clinical and radiographic examination. All implants installed were hollow screw and hollow cylinder implants (Straumann, Waldenburg, Switzerland) with a rough TPS surface. They were placed according to the manufacturer's guidelines. The superstructures consistent in single crowns or fixed partial dentures, which were incorporated 4-6 months postsurgically.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Implant survival rate | 20 years after implants installation

SECONDARY OUTCOMES:
Implant success rate | 20 years after implants installation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Buser, Prof, Study Director — Dep. Oral surgery and Stomatology, University of Bern
Locations (1):
- Chappuis, Bern, Canton of Bern, Switzerland